CLINICAL TRIAL: NCT03366090
Title: Immunological Profiles in Inflammatory Bowel Disease
Acronym: ImmunoIBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Roosenboom, Principal Investigator, Rijnstate Hospital
Other Study IDs: NL62103.091.17
Record Dates: First submitted 2017-06-16; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: IBD; Immunology; Crohn Disease; Ulcerative Colitis; T Cell Subsets; Immunological Profiles
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD patients: Biopsies for immunological analyses
  Interventions: Procedure: Biopsies during coloscopy
- healthy controls: Biopsies for immunological analyses
  Interventions: Procedure: Biopsies during coloscopy

INTERVENTIONS:
Procedure: Biopsies during coloscopy — During standard ileocolonoscopy intestinal biopsy specimens of the macroscopically most inflamed ileal and colonic mucosa will be obtained at the moment of presentation and during follow up.

SUMMARY:
Inflammatory Bowel Diseases (IBD) is a heterogeneous group of diseases regarding clinical presentation, disease course and treatment response. Pathogenesis is complex and multifactorial, based on interactions between genetic and environmental factors, gut microbiota and the immune system, leading to intestinal inflammation. As the immune reaction itself causes the intestinal damage, differences in components of this immune mediated inflammatory reaction between IBD patients might explain the heterogeneity in response to different therapy strategies. Identifying immune components that are associated to disease activity and prognosis would enable a more personalized treatment.

DETAILED DESCRIPTION:
Rationale: Inflammatory Bowel Diseases (IBD) is a heterogeneous group of diseases regarding clinical presentation, disease course and treatment response. Pathogenesis is complex and multifactorial, based on interactions between genetic and environmental factors, gut microbiota and the immune system, leading to intestinal inflammation. As the immune reaction itself causes the intestinal damage, differences in components of this immune mediated inflammatory reaction between IBD patients might explain the heterogeneity in response to different therapy strategies. Identifying immune components that are associated to disease activity and prognosis would enable a more personalized treatment.

Objective: Determine if assessment of mucosal and serological immunological characteristics in combination with clinical indicators of disease behaviour and response to therapy can identify immune-based phenotypes with implications for prognosis and therapeutic interventions.

Study design: The study will be a longitudinal, prospective cohort study. Study population: The study population will include newly diagnosed adults fulling the diagnostic criteria for IBD. These patients will be further studied as a follow up cohort.

Intervention: Immunological analysis of extra mucosal biopsies and venous bloodsamples taken during regular ileocolonoscopy and labcontrols at initial diagnosis and during follow up.

Main study parameters/endpoints: The description of the different mucosal and serological immunological profiles at baseline and follow up in newly diagnosed IBD patients and the correlation between these different immunological profiles and clinical indicators of disease activity, disease course and response to the received therapy.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Ileocolonoscopy with biopsies is a standard examination in patients presenting with chronic (+/- bloody) diarrhoea and in the follow up of patients with IBD. Collection of biopsies during the gastroenterological endoscopy, ie without interventions like polypectomy, is a safe procedure (bleeding, perforation <0,001). In the regular clinical practice, different endoscopists take a variable number of biopsies (4-10) from sites of interest. The intervention in this study comprises taking 4 additional biopsies on top of the regular histological biopsies for immunological examination.

Before ileocolonoscopy, patients normally receive an infusion needle for the administration of sedation (standard care). After ileocolonoscopy this needle will be used to take a venous blood sample. If this is not possible, we take a venous bloodsample during a regular labcontrol. In the follow up period, during regular endoscopies and blood checks the same additional samples will be taken.

Therefore, we believe the burden and risks for patients are minimalised.

ELIGIBILITY:
Inclusion Criteria:

* A patient who meets the following criteria will be included in this study:
* Patients with clinical symptoms of chronic diarrhoea, rectal blood loss, abdominal pain or weight loss who underwent ileocolonoscopy. Macroscopic findings during ileocolonoscopy must suggest IBD, such as erythema, mucosal friability, oedema an bleeding, erosions, superficial or deep ulcerations and luminal narrowing.
* Ultimately, the diagnosis of IBD must be based on a combination of clinical, endoscopic, histologic and radiologic internationally accepted criteria.
* Patients must be able and willing to provide written informed consent.
* Patients above the age of 18, both men and women. AND/OR
* Known IBD patients under treatment during follow up.

Exclusion Criteria:

* A patient who meets any of the following criteria will be excluded from participation in this study:
* Possible new IBD patients who use immunosuppressive medication 4 weeks prior to inclusion (e.g. corticosteroids and anti-TNF therapy) either for IBD, other autoimmune diseases or after organ transplantation.
* Patients diagnosed with an immune suppressive disease.
* Patients who underwent splenectomy in the past.
* Patients diagnosed with any other autoimmune diseases (e.g. Diabetes Mellitus type I, rheumatoid arthritis, celiac disease, psoriasis, systemic lupus erythematosus).
* Patients diagnosed with cancer including hematologic malignancies (e.g. (non-)Hodgkin lymphoma , leukemia), solid tumors and carcinoma in situ, within 5 years before screening with the following caveats:
* Local basal or squamous cell carcinoma of the skin that has been excised and is considered cured is not exclusionary.
* Chronic myelogenous leukemia, hairy cell leukemia, melanoma, renal cell carcinoma, or Kaposi sarcoma are exclusionary irrespective of the duration of time before screening.
* Cervical smear indicating the presence of adenocarcinoma I situ (AIS), high-grade squamous intraepithelial lesions (HSIL), or cervical intraepithelial neoplasia (CIN) of grade>1, is exclusionary, irrespective of the duration of time before screening.
* Follow up IBD-patients who underwent a total colectomy in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include newly diagnosed adults with IBD and the same patients under treatment during follow up.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
The description of the different immunological profiles at baseline and follow up in newly diagnosed IBD patients | 10-2017 till 6-2020
  The description of the different immunological profiles at baseline and follow up in newly diagnosed IBD patients

SECONDARY OUTCOMES:
The correlation between these different immunologic profiles and clinical indicators of disease activity, disease course and response to the received therapy. | 10-2017 till 6-2020
  The correlation between these different immunologic profiles and clinical indicators of disease activity, disease course and response to the received therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No